CLINICAL TRIAL: NCT04214873
Title: A Pilot Study to Evaluate the Effectiveness of the PiQo4 Picosecond Laser (PSL) System for Reduction of Infra-orbital Pigmentation
Brief Title: Evaluation of the Effectiveness of the PiQo4 System for Reduction of Infra-orbital Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Focus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Focus-PiQo4 POH-19-03
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-01

CONDITIONS: POH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- POH (Experimental): Treatment of POH Using PiQo4 Laser System
  Interventions: Device: PiQo4 Laser System

INTERVENTIONS:
Device: PiQo4 Laser System — PiQo4 Laser System for treatment of POH

SUMMARY:
A total of 10 healthy subjects at a single site, aged 18-65 years old and Fitzpatrick skin type I-IV with mild to moderate infra-orbital hyperpigmentation on the background of epidermal and/or dermal pigmentation that wish to improve their POH

ELIGIBILITY:
Inclusion Criteria:

1. Females or males
2. Age 18-65
3. Fitzpatrick skin types I-IV
4. POH on the background of epidermal and/or dermal pigmentation
5. POH severity - mild to moderate
6. Able to read, understand and provide written Informed Consent.
7. Able and willing to comply with the treatment/follow-up schedule and post treatment care
8. Agreed to use the same facial skin care products during the clinical trial period (including the follow-up period)
9. Agreed to the prohibition of the use of local/systemic corticosteroids or retinoids and other local/systemic lightening medications, and willing to abide by such instructions
10. Agreed to the daily use of an over SPF 50 sunblock on their face during the clinical trial period (including the follow-up period), and willing to abide by such instructions
11. Agreed to have their face photographed and willingness to allow Focus Medical (the study Sponsor) and Lumenis and the investigators to use de-identified photographs of the treated area for presentation and publication purposes
12. Women of childrearing potential (not postmenopausal [no menstrual cycle for at least 12 months], without an uterus and/or both ovaries, or has had a bilateral tubal ligation)

    *(In case of women of childbearing potential) Tested negative in the pregnancy test and agreed to use birth control measures during the clinical trial period including use of contraceptives (see list below) IUD, Double-Barrier Method, Vasectomized Partner, No Heterosexual Intercourse, etc
13. Agreed not to undergo any other procedure on their face during their participation in the clinical trial

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Inability to comply with all study protocols and regulations
3. Participation in a study of another device or drug
4. Heavy smokers and/or drinkers (those who smoke 25 or more cigarettes a day and/or ⩾8 drinks a week for women, and ⩾15 for men)
5. Application of any energy device treatment to the infraorbital region within 3 months
6. Application of any dermal filler to the infraorbital region within 6 months
7. Facial resurfacing, deep chemical peels, or taking oral retinoids within 6 months
8. Microdermabrasion (light or medium skin peel) treatment within 30 days
9. Chemical peel, systemic steroids, non-ablative laser, light, or radiofrequency treatment within 3 months
10. Use of topical lightening agents or retinoids within 14 days
11. Any planned surgical intervention to the face for the duration of the trial
12. Use of Latisse, Revitalash, or other lash enhancement stimulators as well as Bimatoprost in the previous 1 month
13. Presence of open wounds, lesions, or scarring in the area
14. Very thin skin (skin that tears, bruises, or breaks easily)
15. Suffering from current or history of significant skin conditions in the treated area that could interfere with the evaluation (i.e. infection, dermatitis, or rash on their face) or requires the use of interfering topical or systemic therapy.
16. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
17. Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex (HSV, HZO) in the treated area, unless treatment is conducted following a prophylactic regimen
18. History of keloid scarring, hypertrophic scarring, or of abnormal wound healing.
19. History of connective tissue diseases such as systemic lupus erythematosus or scleroderma
20. History of post inflammatory pigmentary disorders, particularly a tendency for hyper- or hypo-pigmentation.
21. History of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis.
22. Has used photosensitizing drugs (e.g., Declomycin, sulfa antibiotics, phenothiazines, etc.) within a timeframe where photosensitization from these drugs may still be present
23. History of skin cancer
24. Change of contraceptives dosing in the past 3 months
25. Medical disorders such as thyroid or kidney diseases
26. Significant concurrent illness or any disease state that in the opinion of the Investigator would interfere with the treatment or healing process
27. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Change in POH severity | 3 month follow up
  POH improvement of at least 1 point evaluated by the investigator at the 3-month follow up compared to baseline using the POH severity in comparison to surrounding skin scale where score of between 0 and 4 will be assigned (0-Normal (Skin color comparable to other facial skin areas); 1- Trace (Faint pigmentation of infraorbital fold (bilateral)); 2- Mild (Pigmentation more pronounced); 3- Moderate (Deep dark colour, all four lids involved): ; 4 - Marked (Grade 3 + pigmentation spreading beyond infraorbital fold)

SECONDARY OUTCOMES:
Aesthetic improvement | 3 month follow up
  Aesthetic improvement evaluated by the investigator at the 3-month follow up compared to baseline using a 5-point improvement scale (GAIS) where a score of between 0 and 4 will be assigned (0-Worse (The appearance is worse than the original condition.); 1- No Change (The appearance is essentially the same as the original condition); 2- Improved (Obvious improvement in appearance from initial condition, but a touch-up or re-treatment is indicated.); 3- Much improved (Marked improvement in appearance from initial condition, but not completely optimal. A touch-up would slightly improve the result.); 4 - Very much improved (Optimal result)

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmetic Laser Dermatology, A West Dermatology Company, San Diego, California, United States